CLINICAL TRIAL: NCT05706298
Title: The Effect of Interrupting Sitting With Regular Active Breaks on Glycaemia and Daily Insulin Dose in Sedentary People With Type 1 Diabetes
Brief Title: Active Breaks in People With Type 1 Diabetes
Acronym: EXTOD-Active
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22LJMUSPONSOR010
Record Dates: First submitted 2022-12-21; First posted 2023-01-31 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habitual lifestyle (No Intervention): Participants in the control group will be asked to maintain their habitual lifestyle.
- Active breaks (Experimental): Participants will be asked to interrupt sitting with 3 min bouts of walking every 30 min (16 bouts per day, equalling 48 min of walking) from 9am-5pm every day throughout the 4 week period. To improve adherence should participants miss a bout of walking they will be asked to do 6 min during the next bout.
  Interventions: Behavioral: Active Breaks

INTERVENTIONS:
Behavioral: Active Breaks — Participants will be asked to interrupt sitting with 3 min bouts of walking every 30 min from 9am-5pm
  Arms: Active breaks

SUMMARY:
the investigators aim to determine the effect of 4 weeks of frequent active breaks from prolonged sitting on time in target glycaemic range in people with type 1 diabetes with high habitual sedentary behaviour.

DETAILED DESCRIPTION:
An open-label randomised controlled trial, whereby participants will complete pre-randomisation baseline procedures before allocation to 4wks of habitual activity (control) or active breaks. Interstitial glucose concentrations (fGM), insulin dose and physical activity/ postural transitions (ActivPAL) will be monitored throughout. To improve generalisability and feasibility of recruiting the required number of participants, the study will be completed in a free-living environment using remote data collection methods.

ELIGIBILITY:
Inclusion Criteria:

* T1D diagnosis more than 3 years ago
* Sedentary (> 10h per waking day sedentary (sitting or lying)
* Using insulin therapy with multiple daily injections or insulin pump
* Aged 18-66 (UK retirement age)
* Use of Abbot FreeStyle Libre 2 fGM (>6 weeks to avoid potential lifestyle changes as a result of sensor use)

Exclusion Criteria:

* Engaged in structured planned exercise (e.g. running, cycling, gym, or sports)
* Pregnancy or planning to become pregnant
* <6 months postpartum or stopped breastfeeding <1 month before recruitment
* Existing cerebrovascular or cardiovascular disease
* Significant history of hyperglycaemia (HbA1c >85 mmol/mol)
* History of severe hypoglycaemia requiring third party assistance within the last 3 months

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in time in target glycaemic range | change from baseline to final week of the intervention
  flash glucose monitoring

SECONDARY OUTCOMES:
Change in glycaemic variability (coefficient of variation) | change from baseline to final week of the intervention
  flash glucose monitoring
Change in insulin dose | change from baseline to final week of the intervention
  Insulin dose
Change in Concentration of Hba1c | change from baseline to post intervention (4 weeks)
  HbA1c
Change Insulin to CHO ratio | change from baseline to post intervention (4 weeks)
  Insulin to CHO ratio
Change in Anxiety and depression | change from baseline to post intervention (4 weeks)
  The Hospital Anxiety and Depression Scale (HADS)
Change in Diabetes Quality of Life | change from baseline to post intervention (4 weeks)
  Diabetes Quality of Life (DQOL) questionnaire
Change in Health-related quality of life | change from baseline to post intervention (4 weeks)
  Short Form-12 Health Survey (SF-12)
Change in Height | change from baseline to post intervention (4 weeks)
  Height (cm)
Change in weight | change from baseline to post intervention (4 weeks)
  weight (kg)
Change in BMI | change from baseline to post intervention (4 weeks)
  BMI
Change in waist circumference | change from baseline to post intervention (4 weeks)
  waist circumference (cm)
Change in triglycerides. | change from baseline to post intervention (4 weeks)
  triglycerides.
Change in Insulin Sensitivity Score | change from baseline to post intervention (4 weeks)
  LogeIS
c-peptide | baseline
  c-peptide
Change in sedentary behaviour | change from baseline to final week of the intervention
  minutes of sitting
Change in carbohydrate intake | change from baseline to final week of the intervention
  carbohydrate intake

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jenkins JG, Cocks M, Narendran P, Andrews RC, Shields BM, Scott SN, Lucas SJE, Rendeiro C, Hesketh K. Can 4 weeks of real-world active breaks improve glycaemic management in sedentary adults with type 1 diabetes? The EXTOD-Active randomised control trial protocol. BMJ Open Sport Exerc Med. 2025 Apr 5;11(2):e002594. doi: 10.1136/bmjsem-2025-002594. eCollection 2025. PMID 40195972